CLINICAL TRIAL: NCT04419285
Title: Design of a Mobility Protocol to Assess the Impact of Visual Pathologies in Daily Life Activities for Subjects With Advanced Visual Deficits
Brief Title: Mobility Protocol Adapted for Advanced Visually Impaired Subjects
Acronym: PROMA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier National d'Ophtalmologie des Quinze-Vingts (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: P19-04; 2019-A00937-50 (Other: IDRCB Number)
Record Dates: First submitted 2020-05-07; First posted 2020-06-05 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-04

CONDITIONS: Pigmentary Retinopathy
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Intervention Model Description: The exploratory study will focus on 50 subjects with Retinitis Pigmentosa at very advanced stages
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Retinitis Pigmentosa patients (Experimental): 50 patients with very severe Retinitis Pigmentosa
  Interventions: Behavioral: Locomotion task; Behavioral: Posturology task SOT (Sensory Organization Test); Behavioral: The quality of life questionnaire

INTERVENTIONS:
Behavioral: Locomotion task — The locomotion task takes place on a Streetlab platform. The subject must follow a line on the ground, straight or composed of turns.
  Other Names: Streetlab platform
Behavioral: Posturology task SOT (Sensory Organization Test) — The task takes place on a Streetlab platform with uniform walls without decorations in order to remove any localization element.
  Other Names: Streetlab platform; Opal MobilityLab
Behavioral: The quality of life questionnaire — Study the correlations between the subjects' quality of life scores and the results during behavioral tests. Identify the subjective parameters most sensitive to sensory-motor performance.
  Other Names: NEI-VFQ-25; ULV VFQ (Ultra Low Vision Visual Funnctioning Questionnaire)

SUMMARY:
Retinitis Pigmentosa is characterized by a progressive disappearance of photoreceptors, responsible for a progressive and severe loss of vision.

People Retinitis Pigmentosa therefore encounter a large number of difficulties in daily life, specifically for:

* Visual research
* Visuo-motor coordination in tasks requiring fine motor control
* Visuo-motor coordination in mobility tasks

This study aims to assess the difficulties in the daily life of subjects with Retinitis Pigmentosa at a very advanced stage unsing, quaify of life questionnaires, simplified locomotion tasks in real situation and a posture task.

They are proposing a new test adapted and carried out in real situations, in binocular and monocular vision, making it possible to finely assess locomotion especially for "very low vision" patients.

This test will also ultimately make it possible to better evaluate the effectivements, that is to say to observe and quantify objectively by a score the performance progression obtained for locomotion tasks related to the visual recovery generated by the treatment.

DETAILED DESCRIPTION:
This is monocentric study and the total duration of the study is 48 months. The duration of participation for each research subject is 3 months and maximum 4 visits. This is research involving the human type of non-invasive interventional research, with minimal risks and constraints.

This exploratory study will be conducted on a group of patients with Retinitis Pigmentosa at a very advanced stage.

There will be an inclusion visit including a visual assessment and an ophthalmological consultation. Two experimental visits with tests carried out in a real environment including a locomotion and a posture tasks. An end-of-study visit within a maximum of 1 month following the second experimental visit.

ELIGIBILITY:
Inclusion Criteria:

* Retinitis Pigmentosa, non-syndromic, the diagnosis of which has been confirmed by an ophtmalmologist
* ETDRS visual acuity less than 2/10 (>+0.7 logMAR; <20/100 Snellen)
* Doesn't participate in clinical research that may interfere with this study
* Sufficient knowledge of the French language to ensure a perfect understanding of the tasks to be performed and the instructions received
* Consent to the study signed after information by the investigator
* Health insurance affiliation

Exclusion Criteria:

* Pregnant women
* Inability to give personal consent
* Cataract surgery in the 3 months preceding inclusion
* Amblyopia
* Inability to comply with the instructions for carrying out the study tasks or to complete the study visits
* MMSE score without visual item ≤ 20/25
* Drug treatment which can lead to motor, visual or cognitive disorders (PSA, neuroleptics,etc.) or which may interfere with the study's evaluations

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-03-02 (Actual); Primary Completion 2024-06-02 (Estimated); Study Completion 2024-06-04 (Estimated)

PRIMARY OUTCOMES:
Discriminating | Month 1
  Study of the correlation between the severity of the impairment with regard to visual evaluations (visual acuity, visual field, ect) and the performance score for locomotion and posture tests.
Reproducibility | Month 1
  Graphical and tabular representations will be prepared to represent the correlation between test results and visual function measures on the one hand and daily life activities on the other.
Validity of construction | Month 1
  Graphical and tabular representations will be prepared to represent the correlation between test results and visual function measures on the one hand and daily life activities on the other.

SECONDARY OUTCOMES:
Measurement of postural parameters | Month 1
  The locomotion task which takes place in a Streetlab platform. The subject must follow a line on the ground, straight or composed of turns. For the other tests, the number of turns and the distance to be covered are identical, but the shapes of the courses are systematically different.
  The posturology task SOT (Sensory Organization Test) takes place in a StreetLab platform with uniform walls without decorations so as to remove any localization element.
  The subject is instructed to stand with his hands on his hips as steadily as possible. This test includes 4 experimental conditions for disturbing sensory inputs. the duration of acquisition is 30 seconds, during which the subject must hold a standing position as tatic as possible, without speaking, els hands positioned on the hips while looking straight ahead. Four experimental conditions are tested: Eyes open on a hard floor, eyes closed on a hard floor, eyes open on a foam tray, eyes closed on a foam tray.

CONTACTS AND LOCATIONS:
Overall Officials: Saddek SM MOHAND-SAID, MD, Principal Investigator — Centre Hospitalier National d'Ophtalmologie des Quinze-Vingts
Locations (1):
- Centre Hospitalier National d'Ophtalmologie des Quinze-Vingts, Paris, France